CLINICAL TRIAL: NCT03812328
Title: A Phase 2, Randomized, Active Comparator-Controlled, Open-Label, Adaptive Design Study to Assess the Safety and Efficacy of Intravenously-Administered SelK2 in Patients Undergoing Total Knee Arthroplasty
Brief Title: Study to Assess the Safety and Efficacy of SelK2 to Prevent Blood Clots in Patients Undergoing Total Knee Replacement
Acronym: COURSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tetherex Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SELK2-00005; 2018-003122-88 (EudraCT Number)
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; adhesion molecule; P-selectin glycoprotein ligand 1; P-selectin; venous thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: This was an adaptive design study. The first two arms of the study enrolled patients in a 1:1 ratio to receive either SelK2 or an active comparator. The adaptive arm (SelK2 plus active comparator) was initiated at the discretion of the Steering and Safety Committee. The study then enrolled patients in a 2:1 ratio to receive either SelK2 with an active comparator or an active comparator only.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- SelK2 and Enoxaparin (Experimental): I.V., single-dose (SelK2) and SC, QD for up to 10 ± 2 days (Enoxaparin)
  Interventions: Drug: SelK2; Biological: Enoxaparin
- Enoxaparin (Active Comparator): SC, QD for up to 10 ± 2 days
  Interventions: Biological: Enoxaparin
- SelK2 (Experimental): I.V., single-dose
  Interventions: Drug: SelK2

INTERVENTIONS:
Drug: SelK2 — I.V., single-dose
  Arms: SelK2; SelK2 and Enoxaparin
Biological: Enoxaparin — SC, QD for up to 10 ± 2 days
  Other Names: Lovenox
  Arms: Enoxaparin; SelK2 and Enoxaparin

SUMMARY:
The main purpose of this study is to determine if an investigational medication called SelK2 works in preventing a condition called "venous thromboembolism" (VTE) in patients having a total knee replacement. SelK2 has been designed to attach to a protein found on blood cells and blood vessels. By attaching to this protein, SelK2 is designed to decrease the inflammatory process in the blood vessel wall that leads to the formation of blood clots in the vessel (called thrombosis). By decreasing the inflammatory process, SelK2 may reduce the risk of VTE following joint replacement surgery. In addition, because SelK2 is not a blood thinner, it is expected that the risk for bleeding will also be reduced.

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females, 18-80 years of age (inclusive)
* Planned to undergo elective, primary total unilateral Total Knee Arthroplasty under general anesthesia

Key Exclusion Criteria:

* Previous deep vein thrombosis (DVT) of the leg or pulmonary embolism (PE) within the past year
* Any underlying condition (e.g., atrial fibrillation, mechanical heart valve, or recent pulmonary embolism) that may lead to the required concomitant use of anticoagulants/antiplatelet agents (e.g., warfarin, dabigatran, rivaroxaban, apixaban, clopidogrel) that may affect study outcome or any other drug influencing coagulation (except low dose aspirin (100 mg or less))
* Anticipated use of intermittent pneumatic compression devices and/or electrical/mechanical muscle stimulators post Total Knee Arthroplasty procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Rother, Ph.D., Study Director — Tetherex Pharmaceuticals Corporation
Locations (21):
- Bulgaria (3):
  - UMHAT Kanev AD, Rousse
  - Acibadem City Clinic Tokuda Hospital EAD, Sofia
  - UMHAT Tsaritsa Yoanna - ISUL, Sofia
- Latvia (5):
  - Regional Hospital of Liepaja, Liepāja
  - Hospital of Traumatology and Orthopaedics, Riga
  - ORTO Clinic, Riga
  - Riga's 2nd Hospital, Riga
  - Vidzemes Hospital, Valmiera
- Lithuania (2):
  - Kaunas Clinical Hospital, Kaunas
  - Klaipeda University Hospital, Klaipėda
- Poland (7):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej, Bielsk Podlaski
  - Szpital Ogólny im. dr Witolda Ginela w Grajewie, Grajewo
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow
  - SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodz
  - Wojewódzki Szpital Specjalistyczny, Lublin
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego, Wroclaw
- Ukraine (4):
  - Communal Nonprofit Enterprise Cherkasy Regional Hospital of Cherkasy Oblast Council, Cherkasy
  - Center of Traumatology & Orthopedics, Chernivtsi
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Kiev Regional Clinical Hospital, Kiev

RESULTS

PARTICIPANT FLOW:
Groups:
- Enoxaparin: QD for up to 10 ± 2 days
Period: Overall Study
Arm/Group | SelK2 | SelK2 and Enoxaparin | Enoxaparin
Started | 55 | 63 | 89
Modified Intent-to-Treat (mITT) Population | 48 | 61 | 84
Safety Population | 55 | 63 | 88
Completed | 55 | 60 | 88
Not Completed | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SelK2 | SelK2 and Enoxaparin | Enoxaparin | Total
Number analyzed (Participants) | 55 | 63 | 89 | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 25 | 33 | 78
  >=65 years | 35 | 38 | 56 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (6.35) | 66.3 (7.54) | 65.6 (7.30) | 66.0 (7.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 52 | 68 | 162
  Male | 13 | 11 | 21 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 54 | 63 | 88 | 205
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 55 | 63 | 89 | 207
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Latvia | 15 | 27 | 30 | 72
  Ukraine | 18 | 16 | 27 | 61
  Poland | 11 | 1 | 10 | 22
  Lithuania | 11 | 15 | 18 | 44
  Bulgaria | 0 | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Total Venous Thromboembolism
Description: The primary efficacy endpoint was incidence of total VTE (reported as a percentage of patients) during the Treatment Phase up to venography day (10 ± 2 days after total knee replacement). All efficacy endpoint data was adjudicated by the blinded Central Independent Adjudication Committee (CIAC).
Time Frame: 10 ± 2 Days After Total Knee Replacement
Population: Analysis was performed on the modified intent-to-treat (mITT) population consisting of all randomized patients who also had a successful venogram or symptomatic VTE event, which allowed for assessment of the primary efficacy outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | SelK2 | SelK2 and Enoxaparin | Enoxaparin
Number analyzed (Participants) | 48 | 61 | 84
Participants | 19 | 29 | 17

2. Primary Outcome: Percentage of Participants With Major or Clinically Relevant Non-major Bleeding Events
Description: All suspected bleeding events were reviewed by the Central Independent Adjudication Committee (CIAC) in a blinded fashion and were adjudicated for categorization as Major Bleeding (MB), Clinically Relevant Non-Major Bleeding (CRNMB), Minor Bleeding, or combination of MB and CRNMB. The outcome measure assessed the incidence of MB or CRNMB.
Time Frame: 10 ± 2 Days After Total Knee Replacement
Population: Analysis was performed on the safety population consisting of all patients who received at least 1 dose of study drug, analyzed by actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | SelK2 | SelK2 and Enoxaparin | Enoxaparin
Number analyzed (Participants) | 55 | 63 | 88
Participants | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: Through Day 57
Arm/Group | SelK2 | SelK2 and Enoxaparin | Enoxaparin
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/63 | 0/88
Serious Adverse Events (participants affected / at risk) | 2/55 | 3/63 | 2/88
Other Adverse Events (participants affected / at risk) | 9/55 | 6/63 | 10/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SelK2 (N=55) | SelK2 and Enoxaparin (N=63) | Enoxaparin (N=88)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SelK2 (N=55) | SelK2 and Enoxaparin (N=63) | Enoxaparin (N=88)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 4 (4) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT03812328/Prot_SAP_000.pdf